CLINICAL TRIAL: NCT03195842
Title: Impact of Audio-Recorded Discharge Instructions on Confidence and Comprehension Among Limited English Proficient Parents: A Pilot Randomized Trial
Brief Title: Audio-Recorded Discharge Instructions for LEP Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, K. Casey Lion, Assistant Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00000016
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Limited English Proficiency; Disparities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual discharge care (No Intervention): Standard discharge instructions, meaning conversation with physician, usually via interpreter, along with written instructions compiled by the nurse. Written instructions include pre-translated handouts for common languages, and untranslated (English) patient-specific instructions.
- Recordable card (Experimental): Usual care, as above, plus patient-specific and standard instructions recorded in the patient's preferred language for care and given to them on a card to take home.
  Interventions: Other: Recordable card

INTERVENTIONS:
Other: Recordable card
  Arms: Recordable card

SUMMARY:
In this pilot study, limited English proficient (LEP) parents of children at Seattle Children's Hospital for day surgery will be randomized to usual discharge care or usual discharge plus language-concordant, audio-recorded instructions via recordable card. these cards are similar to recordable greeting cards, and can record up to 180 seconds of information. They can be played back over 100 times. We will follow-up with families 2-7 days later to assess satisfaction and comprehension of discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* Limited English proficient (LEP) parents of day surgery patients at Seattle Children's Hospital (main campus) who prefer one of the following languages for care: Spanish, Somali, Russian, Ukrainian, Vietnamese, Mandarin, or Cantonese. Eligible parents are those receiving condition-specific discharge instructions about one or more of the following: a new medication, wound care, diet advancement, return precautions, or more than 1 follow-up appointment

Exclusion Criteria:

* Child being kept overnight at hospital following surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Comprehension of discharge instructions | 2-7 days after discharge
  Parent-reported instructions (medication, home care, follow-up, and return precautions) compared to documented instructions

SECONDARY OUTCOMES:
Confidence in caring for the child post-discharge | 2-7 days after discharge
  Using 7 health care transition measures
Satisfaction with card | 2-7 days after discharge
  Measures of satisfaction with the recordable card, asked of those who received one

IPD SHARING:
Plan to Share IPD: No